CLINICAL TRIAL: NCT05291624
Title: Concordance Between Ultrasonographic and Surgical Assessment in Patients With Endometriosis by Using AAGL 2021 Endometriosis Classification: a Single-center Prospective Study
Brief Title: Ultrasonographic and Surgical Assessment of Endometriosis by AAGL 2021 Endometriosis Classification
Acronym: ULTRA-AAGL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Piazza della Vittoria 14 Studio Medico - Ginecologia e Ostetricia (Other)
Responsible Party: Principal Investigator, Simone Ferrero, Principal Investigator, Piazza della Vittoria 14 Studio Medico - Ginecologia e Ostetricia
Other Study IDs: ULTRASOUND-AAGL2021
Record Dates: First submitted 2022-03-03; First posted 2022-03-22 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Endometriosis; Bowel Endometriosis; Deep Endometriosis; Ovarian Endometrioma
Keywords: Preoperative Ultrasound; Endometriosis staging; Surgical complexity
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with preoperative suspicion of endometriosis: Consecutive patients undergoing ultrasonographic preoperative assessment and subsequent surgical approach for deep endometriosis
  Interventions: Diagnostic Test: AAGL Endometriosis Classification score - ULTRASOUND; Diagnostic Test: AAGL Endometriosis Classification score - SURGERY

INTERVENTIONS:
Diagnostic Test: AAGL Endometriosis Classification score - ULTRASOUND — At baseline, ultrasonographic evaluation of patients by following AAGL Endometriosis Classification
Diagnostic Test: AAGL Endometriosis Classification score - SURGERY — Within 1 month from enrollment, surgical evaluation of patients by following AAGL Endometriosis Classification

SUMMARY:
In 2021, an international consensus developed a new endometriosis classification system, called AAGL 2021 Endometriosis Classification, for scoring intraoperative surgical complexity and to examine its correlation with patient-reported pain and infertility. Until now, no study has investigated the role of AAGL 2021 Endometriosis Classification in ultrasonographic assessment of patient with endometriosis. This study aims to compare the use of the AAGL 2021 Endometriosis Classification in preoperative (at ultrasound) and intraoperative (at surgery) evaluation of patients with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

- patients with suspected endometriosis undergoing ultrasonographic preoperative evaluation.

Exclusion Criteria:

* patients with suspected or diagnosed malignancy;
* patients a history of colorectal surgery or a surgery for endometriosis including vaginal resection, full-thickness bowel resection or excision of a endometriotic lesion of the urinary bladder;
* patients with previous bilateral ovariectomy.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Patients with suspected endometriosis undergoing ultrasonographic preoperative evaluation and subsequent surgical approach.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Reproducibility between ultrasonographic and surgical AAGL staging (minimum value: 0 points, maximum value: 111 points, higher scores mean a higher surgical complexity) | Through study completion, an average of 1 month
Comparison between total ultrasonographic and surgical AAGL staging score (minimum value: 0 points, maximum value: 111 points, higher scores mean a higher surgical complexity) | Through study completion, an average of 1 month

SECONDARY OUTCOMES:
Comparison between ultrasonographic and surgical AAGL staging subdomains (minimum value: 0 points, maximum value: 111 points, higher scores mean a higher surgical complexity) score | Through study completion, an average of 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Ginecologia - IRCCS Ospedale Sacro Cuore Don Calabria, Negrar, VR, Italy

REFERENCES:
- [Background] Abrao MS, Andres MP, Miller CE, Gingold JA, Rius M, Neto JS, Carmona F. AAGL 2021 Endometriosis Classification: An Anatomy-based Surgical Complexity Score. J Minim Invasive Gynecol. 2021 Nov;28(11):1941-1950.e1. doi: 10.1016/j.jmig.2021.09.709. Epub 2021 Sep 25. PMID 34583009